CLINICAL TRIAL: NCT01606826
Title: Severe Asthma Research Program
Acronym: SARP
Status: Active, not recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Professor of Public Health Sciences, Milton S. Hershey Medical Center
Other Study IDs: SARP003; 1U10HL109086 (NIH); NCT01761058 (obsolete NCT alias)
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Severe
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: CBC/Diff, Total IgE, Serum, Plasma, DNA, RNA; Urine; EBC; Sputum: Supernatant, Cell Pellet; Bronch: BAL, Bronchial Brushings, Bronchial Biopsy
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- Asthmatics: Subjects with active asthma.
- Healthy Controls: Subjects without any known pulmonary disease.

SUMMARY:
The mission of the SARP is to improve the understanding of severe asthma through integrated study of its clinical and biological features and to evaluate their changes over time. The ultimate goal of these efforts is to promote better treatments for severe asthma.

DETAILED DESCRIPTION:
The mission of the SARP is to improve the understanding of severe asthma to develop better treatments. The SARP will gain a better understanding of asthma and its endotypes, in children and adults, by defining the disease at the molecular and cellular levels in the context of the temporal phenotypic expression of the disease. To this end, the SARP investigators will utilize both mechanistic and evoked phenotype approaches to: 1) characterize developmental molecular, cellular and physiologic phenotypes in children and adults with mild to severe asthma, and 2) to further elucidate the evolving pathobiology and pathogenesis of severe asthma and its sub-phenotypes and 3) compare these features over time. This approach involves a shared longitudinal protocol conducted across all participating centers which includes common information on all SARP participants. Additionally, the SARP investigators have each identified mechanistic research questions to be included in the shared longitudinal protocol. Together, these longitudinal and mechanistic approaches will enable prediction of phenotype stability/fluctuation and pharmacologic responses and identification of novel, disease-modifying targets for treatment.

ELIGIBILITY:
Asthmatic Patients:

Inclusion Criteria:

1. Physician diagnosis of asthma,
2. Age 6 years and older
3. Evidence of historical reversibility, including either:

   * FEV1 bronchodilator reversibility ≥ 12%, or
   * Airway hyperresponsiveness reflected by a methacholine PC20 ≤16 mg/mL.

Exclusion Criteria:

1. Pregnancy during the characterization phase,
2. Current smoking,
3. Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age (Note: if a subject has a smoking history, no smoking within the past year),
4. Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion), severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways,
5. History of premature birth before 35 weeks gestation,
6. Unwillingness to receive an intramuscular triamcinolone acetonide injection,
7. Evidence that the participant or family may be unreliable or poorly adherent to their asthma treatment or study procedures,
8. Planning to relocate from the clinical center area before study completion,
9. Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician(s) of record, or
10. Currently participating in an investigational drug trial for asthma therapies.

Healthy Controls:

Inclusion criteria: Healthy subjects between the age of 18 and 65 years. Exclusion criteria

1. History of chronic diseases that affect the lungs,
2. A history suggestive of allergic rhinitis, eczema or chronic sinusitis,
3. An improvement in FEV1 of more than 12% following 4 puffs of albuterol,
4. Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age, or any smoking within the past year,
5. Respiratory tract infection within the past 4 weeks,
6. Pregnancy,
7. History of premature birth (<35 weeks).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target study population will is 80% adults (age 18 and older) and 20% children age 6-17 years, 50% females, and 30% minorities.
  Approximately 100 Healthy Control patients, matching the demographic characteristics of the asthma patients, will also be recruited in order to generate reference data for biospecimens collected from asthmatic patients.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test results | 36 months after enrollment
  Pulmonary function test results include forced expiratory volume in one second (FEV1) and forced vital capacity (FVC).

SECONDARY OUTCOMES:
Frequency of severe asthma exacerbations | 36 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sally Wenzel, MD, Principal Investigator — University of Pittsburgh; Elliot Israel, MD, Principal Investigator — Brigham & Women's Hospital, Boston; Bruce Levy, MD, Study Chair — Brigham & Women's Hospital, Boston; John Fahy, MD, Principal Investigator — University of California, San Francisco; Suzy Comhair, MD, Principal Investigator — The Cleveland Clinic; Loren Denlinger, MD, Principal Investigator — University of Wisconsin, Madison; Wendy Moore, MD, Principal Investigator — Wake Forest University Health Sciences; Mario Castro, MD, Principal Investigator — University of Kansas; David Mauger, PhD, Principal Investigator — Penn State College of Medicine
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Huang BK, Elicker BM, Henry TS, Kallianos KG, Hahn LD, Tang M, Heng F, McCulloch CE, Bhakta NR, Majumdar S, Choi J, Denlinger LC, Fain SB, Hastie AT, Hoffman EA, Israel E, Jarjour NN, Levy BD, Mauger DT, Sumino K, Wenzel SE, Castro M, Woodruff PG, Fahy JV, Sarp FTNSARP. Persistent mucus plugs in proximal airways are consequential for airflow limitation in asthma. JCI Insight. 2024 Feb 8;9(3):e174124. doi: 10.1172/jci.insight.174124. PMID 38127464
- [Derived] Coverstone AM, Boomer JS, Lew D, Bacharier LB, Castro M; Severe Asthma Research Program (SARP) Investigators. Type 2 inflammation in the sputum of adolescents with asthma. Ann Allergy Asthma Immunol. 2021 Mar;126(3):297-299. doi: 10.1016/j.anai.2020.11.018. Epub 2020 Dec 2. No abstract available. PMID 33276117
- [Derived] Ross KR, Gupta R, DeBoer MD, Zein J, Phillips BR, Mauger DT, Li C, Myers RE, Phipatanakul W, Fitzpatrick AM, Ly NP, Bacharier LB, Jackson DJ, Celedon JC, Larkin A, Israel E, Levy B, Fahy JV, Castro M, Bleecker ER, Meyers D, Moore WC, Wenzel SE, Jarjour NN, Erzurum SC, Teague WG, Gaston B. Severe asthma during childhood and adolescence: A longitudinal study. J Allergy Clin Immunol. 2020 Jan;145(1):140-146.e9. doi: 10.1016/j.jaci.2019.09.030. Epub 2019 Oct 14. PMID 31622688
- [Derived] Fitzpatrick AM, Szefler SJ, Mauger DT, Phillips BR, Denlinger LC, Moore WC, Sorkness RL, Wenzel SE, Gergen PJ, Bleecker ER, Castro M, Erzurum SC, Fahy JV, Gaston BM, Israel E, Levy BD, Meyers DA, Teague WG, Bacharier LB, Ly NP, Phipatanakul W, Ross KR, Zein J, Jarjour NN. Development and initial validation of the Asthma Severity Scoring System (ASSESS). J Allergy Clin Immunol. 2020 Jan;145(1):127-139. doi: 10.1016/j.jaci.2019.09.018. Epub 2019 Oct 8. PMID 31604088
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- [Derived] Ricklefs I, Barkas I, Duvall MG, Cernadas M, Grossman NL, Israel E, Bleecker ER, Castro M, Erzurum SC, Fahy JV, Gaston BM, Denlinger LC, Mauger DT, Wenzel SE, Comhair SA, Coverstone AM, Fajt ML, Hastie AT, Johansson MW, Peters MC, Phillips BR, Levy BD; National Heart Lung and Blood Institute's Severe Asthma Research Program-3 Investigators. ALX receptor ligands define a biochemical endotype for severe asthma. JCI Insight. 2017 Jul 20;2(14):e93534. doi: 10.1172/jci.insight.93534. eCollection 2017 Jul 20. PMID 28724795
- [Derived] Phipatanakul W, Mauger DT, Sorkness RL, Gaffin JM, Holguin F, Woodruff PG, Ly NP, Bacharier LB, Bhakta NR, Moore WC, Bleecker ER, Hastie AT, Meyers DA, Castro M, Fahy JV, Fitzpatrick AM, Gaston BM, Jarjour NN, Levy BD, Peters SP, Teague WG, Fajt M, Wenzel SE, Erzurum SC, Israel E; Severe Asthma Research Program. Effects of Age and Disease Severity on Systemic Corticosteroid Responses in Asthma. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1439-1448. doi: 10.1164/rccm.201607-1453OC. PMID 27967215
- See also: Severe Asthma Research Program (SARP) Public Website — http://www.severeasthma.org/